CLINICAL TRIAL: NCT05740917
Title: A Multicenter, Open Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Initial Efficacy of XZB-0004 in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: To Evaluate the Phase I Clinical Study of XZB-0004 in Patients With AML and MDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZB-0004-1002
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: AML; MDS
Keywords: XZB-0004; AXL inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1: XZB-0004 (Experimental)
  Interventions: Drug: XZB-0004

INTERVENTIONS:
Drug: XZB-0004 — XZB-0004 orally Twice daily of every 28-day cycle

SUMMARY:
This is an open-label, multicenter Phase I study that will enroll patients with relapsed/refractory AML or MDS. Stage Ia and stage Ib are included in this study. Phase Ia is a single-agent dose-escalation study that enrolling R/R AML subjects to identify XZB-0004 monotherapy MTD (if any) and RP2D and evaluate its safety and pharmacokinetic profile. Phase Ib will be an expanded study in R/R AML patients (group 1) and R/R MDS patients (group 2) at RP2D doses to further evaluate and determine the efficacy and safety of XZB-0004 in R/R AML or R/R MDS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign written informed consent, able to communicate well with researchers and willing to comply with research regulations.
2. Both men and women can be at least 18 years old at the time of signing the informed consent form.
3. Expected survival ≥ 3 months.
4. The Eastern Cancer Collaboration (ECOG) Physical Fitness score is 0, 1 or 2.

(1) Relapsed or refractory AML that meets the classification criteria of hematopoietic and lymphoid tissue tumors revised by the World Health Organization (WHO) in 2016 and is confirmed by bone marrow cell morphology (except acute promyelocytic leukemia) :

- Criteria for the diagnosis of recurrent AML: recurrence of leukemia cells in peripheral blood after complete response (CR) or ≥5% of primitive cells in bone marrow (except for other causes such as bone marrow regeneration after consolidation chemotherapy) or extramedullary infiltration of leukemia cells.

* Diagnostic criteria for refractory AML:

A) age 18 - 60 one full year of life: Initial treatment cases that did not go into remission after 2 courses of treatment with the standard regimen (containing cytarabine and an anthracycline or anthracquinone); Patients who do not achieve remission after 1 cycle of standard regiments and cannot continue chemotherapy with standard regiments due to age, comorbidities, physical status, and/or adverse risk factors; Or CR after consolidation and intensive treatment, relapse within 12 months; Or recurred 12 months later but failed conventional chemotherapy (no PR or CR); Or two or more relapses; Or extramedullary leukemia persists.

B) Age > 60 years old: Patients who cannot tolerate standard chemotherapy regiments due to age, comorbiditions, physical status, and/or adverse risk factors, or finances were treated with 4 cycles of demethylated drugs (e.g., decitabine or azactidine) and 2 cycles of low-dose chemotherapy ± demethylated drugs.

(2) Relapsed or refractory MDS: Subjects diagnosed by bone marrow cell morphology and cytogenetics WHO (2016) revised classification of MDS as MDS with protocytosis (MDS-EB) :

* Recurrent MDS: Complete response (CR), partial response (PR), or hematological improvement (HI) following at least one of the following responses according to the International Working Group 2006 (IWG 2006) evaluation criteria (see Appendix 7) : ① Bone marrow primitive cells recovered to the pre-treatment level, ② neutrophil absolute count (ANC) or platelet count (PLT) decreased by more than 50% compared with the optimal treatment, ③ hemoglobin (HGB) decreased by more than 15 g/L or depended on blood transfusion;
* Refractory MDS: After adequate treatment (for example, demethylated drug treatment ≥4 cycles), patients meet the criteria of "disease stabilization", "failure", and "disease progression" according to the IWG 2006 efficacy evaluation criteria;
* In addition, if drugs other than methylated drugs progress after treatment or are unable to tolerate toxicity (such as drug-related grade 3 or above liver and kidney toxicity during treatment leading to permanent drug withdrawal); The investigators determined that patients with no other appropriate treatment could also be enrolled.

Stage Ia: meet (1);

Stage Ib Group 1: meet (1);

Stage Ib Group 2: meet (2);

6. Consent for bone marrow aspiration and/or biopsy during screening and treatment.

7. Subject's white blood cell count is less than 30 × 109/L (treatment with hydroxyurea is allowed, but not allowed within 3 days prior to the first treatment with the study drug).

8. Laboratory examination results during the screening period indicate that the subject has appropriate organ function (the following criteria should also be met) :

- Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or endogenous creatinine clearance (CrCl) ≥ 50 mL/min/1.73 m2 as estimated by the Cockcroft-Gault formula (Appendix 2);

* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN (except liver infiltration of leukemia cells);
* Serum total bilirubin (TBIL) ≤ 1.5 ULN (except liver infiltration of leukemia cells);
* Normal or abnormal prothrombin time (PT) and activated partial thrombin time (APTT) had no clinical significance (APTT did not exceed the upper limit of normal for 10s, PT did not exceed the upper limit of normal for 3s);

  9. Women and men of reproductive age must agree, upon signing an informed consent form, to use effective contraceptive methods during the study period and within 6 months after the last dose of XZB-0004.

Exclusion Criteria:

1. Patients with a history of malignancies other than the disease under study within 5 years prior to initial administration of XZB-0004, except those that have been cured for at least 3 years prior to initial administration, such as thyroid carcinoma, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ of the breast, etc.
2. XZB-0004 received systemic antitumor therapy, including chemotherapy, radiotherapy, antibodies, targeted therapy, investigational drugs, etc. within 2 weeks or 5 half-lives prior to initial administration.
3. XZB-0004 was treated with an H2 receptor inhibitor, proton pump inhibitor, or acid suppressor within 3 days prior to initial administration.
4. Adverse reactions caused by previous treatment did not recover to NCI-CTCAE V5.0 level or below (except hair loss and abnormal laboratory examination without clinical significance, etc.).
5. XZB-0004 received adoptive immune cell therapy, including chimeric antigen receptor T cells (CAR), within 12 weeks prior to initial administration.
6. Autologous hematopoietic stem cell transplantation less than half a year, allogeneic hematopoietic stem cell transplantation.
7. Central nervous system leukemia or central nervous system (CNS) invasion.
8. Patients who had received major surgical treatment within 4 weeks prior to the initial administration of XZB-0004.
9. There are serious cardiovascular disease risk factors such as:

   * Chronic heart failure with heart function > Grade 2 (New York Heart Association NYHA scale);
   * If myocardial infarction occurs within 3 months before the first dose, the subject should discuss with the sponsor to confirm his eligibility if his ECG indicates a history of past myocardial infarction;
   * Uncontrolled cardiovascular disease, including unstable angina, clinically uncontrollable hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100 mmHg);
   * Corrected QTcF interval using Fridericia's formula (Appendix 2); 450msec (male) and > 470msec (female).
   * Left ventricular ejection fraction (LVEF) < 50%
10. Active infection is present.
11. Inability to take medications orally.
12. Suffering from active peptic ulcer, Crohn's disease, apparent vomiting, chronic diarrhea, intestinal obstruction, malabsorption, or other diseases known to affect drug absorption; Having difficulty swallowing or other conditions that severely affect drug absorption, such as having undergone a gastrectomy or enterectomy.
13. Active hepatitis B (HBsAg and/or HBcAb positive with HBV-DNA > 500IU/mL) or hepatitis C virus infection (anti-HCV positive with HCV-RNA positive) or human immunodeficiency virus (HIV) antibody positive or syphilis antibody positive.
14. Pregnant or lactating women.
15. There are other severe, acute or chronic medical or mental illnesses or laboratory abnormalities that, in the judgment of the investigator, may increase the risks associated with study participation or may interfere with the interpretation of the findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (for Part 1) | 28 days following first dose of XZB-0004
  Determine MTD of XZB-0004
Overall Response Rate (ORR) (for Part 2) | 2 years after first dose of XZB-0004
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1.

SECONDARY OUTCOMES:
Area under the concentration versus time curve of XZB-0004 in plasma (AUC) | 2 months after first dose of XZB-0004
  To determine the area under the plasma concentration time curve (AUC) of XZB-0004
Maximum plasma concentration (Cmax) of XZB-0004 | 2 months after first dose of XZB-0004
  Cmax is the maximum observed plasma concentration in ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China